CLINICAL TRIAL: NCT05071560
Title: Pilot Study of Supervised Adapted Physical Exercise in Women With Breast Cancer After Treatment - Face-to-face Context vs Online Home Based
Brief Title: Physical Exercise for Breast Cancer Survivors: Face-to-face Versus Home-based
Acronym: On4Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Universidad Europea de Madrid (Other); University Institute of Maia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: On4Rehab Pilot Trial
Record Dates: First submitted 2021-07-04; First posted 2021-10-08 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face Group (Active Comparator): This arm will have a 3 day per week face-to-face participant-tailored combined exercise program, with 2 supervised sessions and 1 non supervised aerobic session, for 8 weeks
  Interventions: Other: Combined exercise training
- Home-Based Group (Experimental): This arm will have a 3 day per week home-based participant-tailored combined exercise program, with 2 remotely supervised sessions (online) and 1 non supervised aerobic session, for 8 weeks
  Interventions: Other: Combined exercise training

INTERVENTIONS:
Other: Combined exercise training — Before the intervention, these women will undergo an evaluation of cardiorespiratory fitness, functional fitness, psychological status and a physiatry assessment. A consent form is signed before the start.
  The physical exercise intervention was planned based on the recommendations of the American College of Sports Medicine for cancer survivors (ACSM 2019), with two supervised combined training sessions (mobility, aerobic training, strength and flexibility training) planned, and one unsupervised aerobic training session per week, interspersed with at least one rest day in between, for 8 weeks. The intensity will be individualized and defined based on the initial assessment. The structure of the training plan was based on the FITT-VP principles (frequency, intensity, time, type, volume and progression) recommended by the ACSM (2019).

SUMMARY:
The present investigation is a pilot feasibility study that aims to compare a physical exercise intervention in a face-to-face context (considered state of the art) with a physical exercise intervention in a distance context (online), both supervised, in women, of legal age, physically inactive, breast cancer survivors after primary treatment with curative intent.

Before and after the intervention these women will have a physical and functional assessment, as well as a pre-trial cardiopulmonary exercise test, to check if there are safety conditions to participate and also to self tailor the exercise prescription.

The prescription follows the ACSM´s exercise guidelines for cancer survivors and will comprise a 8 week combined exercise training, 3 times per week, in which two of them will be supervised and the third session of the week (cardio session) won´t.

Chat´s and weekly personal messages, as well as education, will be used to promote retention and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Over legal age
* With diagnosis of breast carcinoma between stages 0 and IIIc
* ECOG 0 to 1
* Undergoing primary treatment with curative intent (surgery associated or not, with chemotherapy and / or adjuvant radiotherapy) for at least one month
* With follow-up on medical oncology consultation at CHVNG/E
* With consent of the attending oncologist for the practice of physical exercise
* Non-compliance with current physical activity guidelines recommended by the ACSM (moderate aerobic activity> = 150 min / week or vigorous> = 75 min / week and > = 2 strength training sessions / week)
* With cognitive capacity to understand the project proposal

Exclusion Criteria:

* Severe anaemia seen in the last 3 months (Hb <= 8g / dl) or moderate (Hb> 8 and <= 10 g / dl) symptomatic (sustained tachycardia, exertional dyspnea, chest pain or syncope),
* Uncontrolled arterial hypertension (HTN grade 3-4 (CTCAE v.5)) (SAD> = 160mmHg and / or DAD> = 100mmHg) and / or potentially fatal consequences (malignant HTN, transient or permanent neurological deficit or hypertensive crisis)
* Uncontrolled diabetes mellitus
* Known cardiac or respiratory pathology
* Any other contraindication given by the physiatrist and / or assistant surgeon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Retention rate | End of the intervention (week 9)
  The percentage of included patients who ended the program
Adherence rate | End of the intervention (week 9)
  Number of absences to the sessions and number of completed sessions
Training tolerance regarding the duration of the exercise prescription | During all intervention sessions (24 sessions, 8 weeks)
  Recording adherence to the exercise prescription duration, possible adjustments and their reasons
Training tolerance regarding the intensity of the exercise prescription | During all intervention sessions (24 sessions, 8 weeks)
  Recording adherence to the exercise prescription intensity, possible adjustments and their reasons
Training tolerance regarding the volume of the exercise prescription | During all intervention sessions (24 sessions, 8 weeks)
  Recording adherence to the exercise prescription volume, possible adjustments and their reasons
Intervention Recruitment Rate | Beginning of the intervention (week 0)
  Number of invitations made versus accepted (invitation made by the assistant oncologist)
Training safety | During all intervention sessions (24 sessions, 8 weeks)
  Recording symptoms and adverse effects
Absence and dropout | End of the intervention (week 9)
  Rate of absence from sessions and dropout of the program
Level of satisfaction | End of the intervention (week 9)
  Questionnaire at the end of the intervention, from 1 to 5, where 1 is not satisfied and 5 is very satisfied

SECONDARY OUTCOMES:
Cardiopulmonary system fitness level and signs of disease assessment | Beginning of the intervention (week 0)
  Measurement of maximum VO2 by a cardiopulmonary exercise test and assessment of cardiopulmonary risk factors or disease
Lower limb strength | Beginning (week 0) and End of the intervention (week 9)
  30´´Sit to stand test (number of repetitions)
Upper limb strenght | Beginning (week 0) and End of the intervention (week 9)
  Bilateral handgrip test with dynamometer (kg)
Lower limbs flexibility level | Beginning (week 0) and End of the intervention (week 9)
  Sit and Reach test (cm)
Static balance | Beginning (week 0) and End of the intervention (week 9)
  One Leg Stance test (time, s)
Dynamic balance and agility | Beginning (week 0) and End of the intervention (week 9)
  8 Foot up and go test (time, s)
Assessment of aerobic capacity | Beginning (week 0) and End of the intervention (week 9)
  6 Minute Walk Test
Safety of the intervention | During all intervention sessions (24 sessions, 8 weeks)
  Number of serious and less serious occurrences
Body weight | Beginning (week 0) and End of the intervention (week 9)
  Weight (Kg)
Body height | Beginning (week 0) and End of the intervention (week 9)
  Height (m)
Body circumferences | Beginning (week 0) and End of the intervention (week 9)
  Waist circumference (cm), hip circumference (cm), middle crural circumference (cm) and bicipital circumference (cm)
Individual's overall satisfaction with life and general sense of personal well-being | Beginning (week 0) and End of the intervention (week 9)
  Questionnaire QLQ-C30
Individual's overall satisfaction with life and general sense of personal well-being, specific to breast cancer patient | Beginning (week 0) and End of the intervention (week 9)
  Questionnaire QLQ-BR23
Adverse effects | During all intervention sessions (24 sessions, 8 weeks)
  Common Terminology Criteria for Adverse Effects, version 5, scale (presence of fatigue, osteoarticular and cardiac complaints, pain, neuropathy and lymphedema), ranging from 1 (mild, asymptomatic ou mild symptoms) to 5 (dead related to adverse event)
Assessment of performance status | During all intervention sessions (24 sessions, 8 weeks)
  ECOG scale of performance status, in a scale ranging from 0 (fully active, able to carry same activities as before disease without new restrictions) to 5 (dead)
Heart Function | Beginning of the intervention (week 0)
  Resting heart rate (bpm)
Arterial disorder assessment | Beginning of the intervention (week 0)
  Systolic and diastolic blood pressure assessment (mm/hg)
Physical activity and sedentary behaviors | Beginning (week 0) and End of the intervention (week 9)
  Accelerometry
Subjective perception of effort | During all intervention sessions (24 sessions, 8 weeks)
  Borg scale of perceived exertion ranging from 6 (very, very light effort) to 20 (maximum exertion)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Martins, PhD, Study Director — Universidade Europeia
Locations (1):
- Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be available with the exception of personal information
Supporting Information: Study Protocol, SAP, ICF, CSR